CLINICAL TRIAL: NCT06075602
Title: COMPLEX Registry - a Prospective COhort Study to Describe the Management and Outcomes of Patients Presenting with CompLEX and Calcified Coronary Artery Disease
Acronym: COMPLEX
Status: Recruiting | Type: Observational
Sponsor: Luzerner Kantonsspital (Other)
Responsible Party: Principal Investigator, Matthias Bossard, Principal Co-Investigator, Luzerner Kantonsspital
Other Study IDs: 2021-01290
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Coronary Disease; Coronary Artery Disease; Coronary Restenosis; Coronary Arteriosclerosis; Coronary Artery Calcification; Stable Chronic Angina; Angina Pectoris; Angina, Stable; Angina, Unstable; Stent Thrombosis
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease; Coronary Restenosis; Angina, Stable; Angina Pectoris; Angina, Unstable | interventions — Equipment and Supplies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Treatment: The project ́s main goal is to collect baseline, clinical and procedural data as well as to assess angiographic and clinical outcomes of patients with complex coronary lesions treated with current PCI techniques/ devices, but also CABG strategies in different clinical settings.
  Interventions: Device: Impact of current PCI techniques/ devices in complex coronary artery lesions

INTERVENTIONS:
Device: Impact of current PCI techniques/ devices in complex coronary artery lesions — To evaluate the impact of current PCI techniques/devices, but also CABG strategies, in patients with complex coronary artery lesions

SUMMARY:
The purpose of the COMPLEX Registry is to prospectively and retrospectively collect baseline, clinical and procedural data of patients who have undergone PCI or CABG for complex and/ or calcified chronic CAD, irrespective of clinical presentation as well as to prospectively collect data about their clinical outcomes. The outcomes will be compared in different clinical subgroups (e.g. PCI vs. CABG). The impact of current PCI techniques/ devices, but also CABG strategies in different clinical settings and coronary artery lesions on cardiovascular outcomes will be assessed.

DETAILED DESCRIPTION:
a. PCI cohort - Periprocedural outcomes/ complications to be analyzed represent: final result (e.g. TIMI flow), stent expansion, dissections, perforations, and prevalence of thrombus (assessed by angiography and intravascular imaging) b. CABG cohort - Periprocedural outcomes/ complications to be analyzed include: final result (e.g. graft flow), number and type of grafts, total length of surgery, bypass time, cross-clamp time, median chest-tube output (mL), bleeding, duration of CCU/ ICU stay, re-operation.

c. For the PCI, CABG as well as medically managed cohort, short and long-term clinical outcomes of interest include: unstable angina (UA), stent-/scaffold thrombosis, target lesion failure (TLF), target vessel revascularization (TVR), ischemia driven revascularization, repeat hospitalization, new/worsening heart failure, cardiogenic shock, stroke, bleedings, cardiovascular death and all-cause death.

2. PCI cohort:

1. To describe procedural and clinical performance of various PCI devices including high pressure balloons, scoring, balloons, cutting balloons, rotational atherectomy, orbital atherectomy, intravascular lithotripsy, stent and scaffold devices implanted in patients presenting with complex and calcified chronic CAD
2. To study the impact of different PCI devices and revascularization strategies used for lesion preparation and PCI optimization strategies among patients undergoing PCI
3. To describe early and late angiographic and OCT-findings among complex and calcified coronary artery disease patients treated with various metallic stent and scaffold devices
4. To assess possible predictors for coronary stent implantation or device failure 3. CABG cohort:

a. To describe procedural and clinical performance of various surgical techniques b. To assess outcomes across various surgical cohorts (e.g. urgent vs. elective, diabetic vs. non-diabetic, gender disparities) c. To investigate various CABG revascularization strategies (e.g. off- versus on-pump, "Fully arterial", minimal invasive approach) and their impact on short and long-term outcomes d. To describe perioperative recovery and risk for in-hospital complications (e.g. wound infections, pneumonia) e. To assess possible predictors for graft failure with contemporary surgical techniques 4. Conservative - only medically treated - cohort:

1. To describe medical management (drugs regimens) as well as other lifestyle interventions in patients presenting with complex and calcified chronic CAD who are being treated with a primarily conservative (non-invasive) strategy.
2. To study the clinical impact of different treatment strategies/ medical regimens used among chronic, complex CAD, which are being managed solely with medical therapy.
3. To assess possible predictors for management failure (e.g. recurrence of symptoms or impaired quality of life).

   5. To compare presentation, (medical) management, short- and long-term outcomes across the different treatment cohorts (PCI, CABG and medically managed cohort).

   6. To specifically describe age- and gender-specific disparities across the various treatment regimens (e.g. PCI versus CABG).

   7. To evaluate the impact of different antithrombotic regimens on patient's clinical outcomes 8. To study procedural and clinical outcomes among CAD patients requiring hemodynamic support using mechanical devices.

   9. To analyze the performance of various non-invasive testing modalities (e.g. laboratory/ ECG parameters, treadmill-test, stress-echocardiography, CMR, SPECT or PET-CT) in order to predict outcomes of patients with chronic, complex CAD.

   10. To describe economic implications (cost-effectiveness) of various interventional treatments for CAD.

ELIGIBILITY:
Inclusion Criteria:

* Subject >18 years of age
* Individuals presenting with chronic, complex and/or calcified CAD and requiring PCI or CABG
* Complex coronary artery disease / lesions must include at least one of the following attributes:
* Long and/ or heavily calcified coronary lesions
* In-stent restenosis
* Chronic total occlusions (CTO)
* Left main lesions
* Bifurcation lesions
* Bypass graft lesions
* Small vessel disease / coronary microvascular dysfunction (e.g. not amenable to PCI)
* Subjects must be willing to sign a patient informed consent (PIC) or must have signed the General Consent (GK).

Exclusion Criteria:

The presence of any one of the following exclusion criteria will lead to exclusion of the patient.

* Patient is <18 years of age
* Patient unwilling or unable to provide informed consent
* Patients with no complex and calcified CAD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In an all-comers design, virtually any CAD patient with complex and/ or calcified coronary artery disease treated with PCI or CABG at the Heart Center of the Luzerner Kantonsspital (LUKS) and giving consent may be included.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Major adverse cardiac and cerebrovascular events (MACCE) | 1 year

SECONDARY OUTCOMES:
Rate of combination of major adverse cardiac and cerebrovascular events (MACCE) | 1 year, 2 years, 5 years and 10 years
Rate of acute vessel closure | 1 year, 2 years, 5 years and 10 years
Rate of target vessel revascularization (TVR) | 1 year, 2 years, 5 years and 10 years
Rate of target lesion revascularization (TLR) | 1 year, 2 years, 5 years and 10 years
Rate of target lesion failure (TLF) | 1 year, 2 years, 5 years and 10 years
Rate of ischemia driven TLR | 1 year, 2 years, 5 years and 10 years
Rate of new AMI (NSTEMI/STEMI) | 1 year, 2 years, 5 years and 10 years
Rate of TIA or stroke | 1 year, 2 years, 5 years and 10 years
Rate of cardiovascular mortality | 1 year, 2 years, 5 years and 10 years
Rate of all-cause mortality | 1 year, 2 years, 5 years and 10 years
Rate of bleeding events (access site or non-access site related) according to the BARC classification. | 1 year, 2 years, 5 years and 10 years
Rate of vascular complications (according to VARC criteria) | 1 year, 2 years, 5 years and 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Florim Cuculi, MD, Principal Investigator — Luzerner Kantonsspital
Locations (1):
- Lucerne Heart Centre, Lucerne, Canton of Lucerne, Switzerland

REFERENCES:
- [Background] Seiler T, Attinger-Toller A, Cioffi GM, Madanchi M, Teufer M, Wolfrum M, Moccetti F, Toggweiler S, Kobza R, Bossard M, Cuculi F. Treatment of In-Stent Restenosis Using a Dedicated Super High-Pressure Balloon. Cardiovasc Revasc Med. 2023 Jan;46:29-35. doi: 10.1016/j.carrev.2022.08.018. Epub 2022 Aug 20. PMID 36085285
- [Background] Madanchi M, Cioffi GM, Attinger-Toller A, Wolfrum M, Moccetti F, Seiler T, Vercelli L, Burkart P, Toggweiler S, Kobza R, Bossard M, Cuculi F. Long-term outcomes after treatment of in-stent restenosis using the Absorb everolimus-eluting bioresorbable scaffold. Open Heart. 2021 Sep;8(2):e001776. doi: 10.1136/openhrt-2021-001776. PMID 34518287
- [Background] Pinilla-Echeverri N, Bossard M, Hillani A, Chavarria JA, Cioffi GM, Dutra G, Guerrero F, Madanchi M, Attinger A, Kossmann E, Sibbald M, Cuculi F, Sheth T. Treatment of Calcified Lesions Using a Dedicated Super-High Pressure Balloon: Multicenter Optical Coherence Tomography Registry. Cardiovasc Revasc Med. 2023 Jul;52:49-58. doi: 10.1016/j.carrev.2023.02.020. Epub 2023 Mar 2. PMID 36907698
- [Background] Madanchi M, Cioffi GM, Kobza R, Cuculi F, Bossard M. The Importance of Defining the Coronary Anatomy in Suspected Myopericarditis: A Case Report. Am J Case Rep. 2021 Mar 29;22:e929009. doi: 10.12659/AJCR.929009. PMID 33780431
- [Background] Bossard M, Madanchi M, Avdijaj D, Attinger-Toller A, Cioffi GM, Seiler T, Tersalvi G, Kobza R, Schupfer G, Cuculi F. Long-Term Outcomes After Implantation of Magnesium-Based Bioresorbable Scaffolds-Insights From an All-Comer Registry. Front Cardiovasc Med. 2022 Apr 14;9:856930. doi: 10.3389/fcvm.2022.856930. eCollection 2022. PMID 35498044